CLINICAL TRIAL: NCT05427994
Title: Assessing the Quality of Life and Social Support in Age-Related Macular Degeneration Patients
Status: Completed | Type: Observational
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Ildar Fakhradiyev, Principal Investigator, Asfendiyarov Kazakh National Medical University
Other Study IDs: 1394
Record Dates: First submitted 2022-06-15; First posted 2022-06-22 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Age-Related Macular Degeneration
Keywords: age-related macular degeneration; quality of life; social support; reliability of social support; vision related quality of life
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with age-related macular degeneration: Patients with age-related macular degeneration who fill out the quality of life questionnaire, and answer questions about social support and reliability of social support
  Interventions: Other: National Eye Institute Visual Function Questionnaire

INTERVENTIONS:
Other: National Eye Institute Visual Function Questionnaire — National Eye Institute Visual Function Questionnaire (NEI-VFQ-25) measures the quality of life related to vision. This questionnaire has been validated for use on low vision patients.
  Other Names: NEI-VFQ-25

SUMMARY:
The aim of this study is to evaluate the quality of life of AMD patients related to vision using the short version of the National Eye Institute Visual Function Questionnaire (NEI-VFQ-25), patients' social support, and their relationship with demographic and clinical variables.

DETAILED DESCRIPTION:
Background and study aims. Age-related macular degeneration (AMD) is the most prevalent chronic progressive ocular disease. It has been shown in several studies that AMD affects the quality of life of patients. The aim of this study is to evaluate the quality of life of AMD patients related to vision using the short version of the National Eye Institute Visual Function Questionnaire (NEI-VFQ-25), patients' social support, and their relationship with demographic and clinical variables.

Who can participate? Patients with AMD, who wish to participate, will be recruited. Patients will be recruited from three locations of the Kazakh Scientific - Research Institute of Eye Diseases in Almaty, Nur-Sultan and Shymkent.

What does the study involve? The study involves collecting demographic data of the participants, collecting baseline visual testing data from medical records, filling out of the NEI-VFQ-25, and answering two yes/no questions related to the social support and reliability of social support.

What are possible benefits and risks of participating? Assessment of quality of life and social support of the AMD patients is a first step of developing targeted psycho-social support programs for AMD patients.

Where is the study run from? Patients will be recruited from three locations of the Kazakh Scientific - Research Institute of Eye Diseases in Almaty, Nur-Sultan and Shymkent.

When is the study starting and how long it is expected to run for? Start date 03/02/2020. End date 27/08/2022.

Who is funding the study? No funding for this study. Who is the main contact? Principal investigator: Inara Ismailova; +380 73 200 0688; i.ismayilova@gmail.com

ELIGIBILITY:
Inclusion Criteria:

* age-related macular degeneration; ability to speak and understand Russian and/or Kazakh language; willingness to participate

Exclusion Criteria:

* Presence of glaucoma, cataracts of grade 2 or more according to the Lens Opacities Classification System (LOCS) III, and the presence of corneal opacities or any other retinal diseases

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed age-related macular degeneration
Sampling Method: Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Quality of life of AMD patients | at the recruitment to the study
  Vision related Quality of life (QOL) of AMD patients related to vision assessed by NEI-VFQ-25 total score at the recruitment. NEI-VFQ-25 has 38 questions with multiple choice answers, each rated 0,25, 50, 75 or 100. The overall score is measured as a mean of all answers

SECONDARY OUTCOMES:
Social Support | at the recruitment to the study
  Percentage of AMD patients with Social Support. Social Support of AMD patients at the recruitment assessed by answering a yes/no question.
Reliability of Social Support | at the recruitment to the study
  Percentage of AMD patients with a reliable Social Support. Reliability of Social Support of AMD patients at the recruitment assessed by answering a yes/no question.
Relationship between QOL and social support | at the recruitment to the study
  Correlation between the overall quality of life of AMD patients and demographic, visual characteristics, and social support tested with multiple linear regression model. The Hosmer-Lemeshow goodness-of-fit test will be used to test the model's fit. All tests will be two-tailed with a significance level of 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Inara Isamyilova, PhD, Principal Investigator — Asfendiyarov Kazakh National Medical University
Locations (2):
- Kazakhstan (2):
  - Kazakh Scientific - Research Institute of Eye Diseases, Almaty
  - Medical Centre Hospital of President'S Affairs Administration of the Republic of Kazakhstan, Astana

IPD SHARING:
Plan to Share IPD: No
According to the patient consent form data is not available for scientific use by others than the project group members.

REFERENCES:
- [Derived] Ismayilova I, Turdaliyeva B, Aldasheva N, Veselovskaya N. Assessing the quality of life in age-related macular degeneration patients: a cross-sectional study in Kazakhstan. Acta Biomed. 2022 Dec 16;93(6):e2022299. doi: 10.23750/abm.v93i6.13580. PMID 36533748